CLINICAL TRIAL: NCT04621357
Title: Consequences of Oedema on the Prognosis of InTraCerebral Haemorrhage
Brief Title: Influence of Cerebral Oedema in Intracerebral Haemorrhage
Acronym: COPITCH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Conseil Régional Hauts-de-France, France (Unknown); Fondation pour la recherche sur les AVC (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017_70; 2019-A02502-55 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2020-10-29; First posted 2020-11-09 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Stroke; Intra Cerebral Hemorrhage
Keywords: Intra Cerebral Hemorrhage; Perihaematomal oedema; MRI; outcome
MeSH Terms: conditions — Stroke; Cerebral Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patient with intracerebral haemorrhage (Experimental): Patients will be screened at admission in the stroke units right after brain MRI demonstrating the presence of blood in the brain parenchyma.
  Interventions: Radiation: Brain MRI; Biological: Biological biomarkers

INTERVENTIONS:
Radiation: Brain MRI — Brain MRI will include differents sequences.
Biological: Biological biomarkers — Biological biomarkers will include a set of systemic inflammatory markers

SUMMARY:
In 2020, IntraCerebral Haemorraghe (ICH) remains the most devastating type of stroke. Besides stroke unit care, no specific treatment has been proven effective yet. Perihaematomal oedema (PHO) could be a promising therapeutic target. However, the mechanisms, the natural history as well as the clinical impact of this PHO remain unclear. The COPITCH study has been designed to answer these questions

ELIGIBILITY:
Inclusion Criteria:

* With a spontaneous ICH, i.e. non traumatic
* Admitted within 12 hours of stroke onset. For wake-up strokes, time of last seen well will be considered as stroke onset
* Patient insured under the French social security
* Consent form signed

Exclusion Criteria:

* Pure intraventricular haemorrhages
* "secondary" ICH: ICH resulting from intracranial vascular malformation, intracranial venous thrombosis, head trauma or tumour; haemorrhagic transformation within an infarct
* Pre-admission modified Rankin score of 4 or 5
* Life expectancy of less than 1 year related to comorbidities (end stage cancer, end stage organ failure)
* Pregnancy or breastfeeding or Women of childbearing age without effective contraception (a pregnancy test will be done)
* Adults who are deprived of their liberty by judicial or administrative decision
* Referral from other hospitals
* Contra-indication to MRI : claustrophobia, ocular metallic foreign bodies (accidental or other) or in a risk area (nervous or vascular system);irremovable implanted medical device (pacemaker, neurostimulator, cochlear implants and others);metallic heart valve (mainly old heart valves) or vascular clips previously implanted on cranial aneurysms; gadolinium allergy
* No consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2021-06-04 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Poor functional outcome defined as a modified Rankin Scale of 4 or more | at 3 months

SECONDARY OUTCOMES:
overall distribution of the modified Rankin scale at 3- and 12 months | at 3 months and 12 months
  The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability.
  The scale runs from 0-6, running from perfect health without symptoms to death.
Early neurological deterioration defined as more than 4 points on the NIHSS score | at 96 hours
  The NIHSS score (NIH Stroke Scale) is used to monitor the progression of an ischemic or hemorrhagic stroke. It is rated from 0 to 42 points. Depending on the result, a distinction is made from Minor stroke to Severe stroke
all-cause mortality at 3 and 12 months | at 3 and 12 months
Cognitive decline | at 3 months, at 12 months
  Cognitive decline defined as a score on MOCA test below 27

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Cordonnier, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- CHU de Lille, Lille, France